CLINICAL TRIAL: NCT07186738
Title: Study of a Patient Cohort Following Digestive Surgical Care After the Implementation of a Telemonitoring and Tele-coordination Platform for Medical, Paramedical, and Social Management
Acronym: EPOCA
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Principal Investigator, bp-prom-regl, MD PhD, Nantes University Hospital
Other Study IDs: AP_ED_EPOCA
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Telemonitoring
Keywords: telemonitoring; digestive surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- telemonitoring patient after digestive surgery: EPOCA telemonitoring at home for patients following digestive surgery
  Interventions: Device: EPOCA telemonitoring

INTERVENTIONS:
Device: EPOCA telemonitoring — EPOCA is a telemonitoring and tele-coordination platform for medical, paramedical, and social care, enabling the follow-up of acute or chronic patients at home-whether after hospital discharge, as an alternative to hospitalization, or for long-term monitoring. The EPOCA solution relies on connected devices, a digital platform for analyzing incoming data, and a team of medical and paramedical professionals for monitoring and coordination. Remote medical monitoring includes teleconsultations, at-home paramedical care, guidance and support for families, nursing homes, or long-term care facilities, and 24/7 management of home emergencies

SUMMARY:
Postoperative hospital stays and complications vary widely after digestive surgery. Enhanced Recovery After Surgery (ERAS) protocols have shortened stays and accelerated recovery after elective procedures, but they remain challenging in emergency surgery and among frail or elderly patients. While theoretical discharge after colorectal surgery is possible between postoperative days 2 and 7, average stays in practice are 12-14 days. Bariatric surgery similarly targets discharge on days 2-3, yet typical stays are 8-10 days. Patients successfully managed under ERAS may face higher readmission risk, often due to worsening comorbidities or serious complications.

Prolonged hospitalization and readmissions impact patient safety, comfort, and healthcare costs. Daily hospital costs in surgical units range from €350 to €400. Post-acute care facilities can reduce readmissions but often have long waiting periods. To minimize readmission risk, many surgeons prefer in-hospital postoperative monitoring, limiting early discharge.

Recent studies show that connected devices and teleconsultation can provide safe and effective postoperative follow-up. Teleconsultation follow-up is feasible for most patients, with satisfaction rates comparable to in-person visits. Remote monitoring of stoma care has been associated with reduced readmissions. Home-based monitoring using connected vital sign devices in high-risk patients reduces readmissions and emergency visits. In colorectal and bariatric surgery, daily remote monitoring after early discharge (24-48 hours) did not increase morbidity or readmission, suggesting that telemonitoring can safely enable earlier discharge while maintaining patient safety. Continuous monitoring is particularly important for high-risk patients due to rapid deterioration from potential complications.

EPOCA is a telemonitoring and telecoordination platform providing medical, paramedical, and social follow-up at home. It combines connected devices, a digital platform for data analysis, and a dedicated medical and paramedical team. Services include teleconsultations, home paramedical care, support for families or care facilities, and 24/7 emergency management.

EPOCA reassures patients and caregivers, supports primary care and home care teams, and integrates hospital and emergency services. It addresses challenges posed by aging populations, chronic disease prevalence, and increasingly complex patients. By enabling earlier discharge without increasing readmissions, EPOCA offers a holistic solution bridging hospital and home care. It has already demonstrated success in preventing hospitalizations in high-risk elderly patients and is authorized for telemonitoring of chronic conditions including diabetes, respiratory, renal, and cardiac insufficiency.

This study aims to evaluate the feasibility of implementing EPOCA over two years in the CHU Nantes digestive surgery unit. It will target patients undergoing elective or urgent colorectal or bariatric surgery who are at risk of prolonged hospitalization or readmission. High-risk scenarios include anticipated early discharge within 24 hours and patients identified as having elevated readmission risk according to predefined criteria

DETAILED DESCRIPTION:
Postoperative hospital stays and complications vary widely after digestive surgery. Enhanced Recovery After Surgery (ERAS) protocols have shortened stays and accelerated recovery after elective procedures, but they remain challenging in emergency surgery and among frail or elderly patients. While theoretical discharge after colorectal surgery is possible between postoperative days 2 and 7, average stays in practice are 12-14 days. Bariatric surgery similarly targets discharge on days 2-3, yet typical stays are 8-10 days. Patients successfully managed under ERAS may face higher readmission risk, often due to worsening comorbidities or serious complications.

Prolonged hospitalization and readmissions impact patient safety, comfort, and healthcare costs. Daily hospital costs in surgical units range from €350 to €400. Post-acute care facilities can reduce readmissions but often have long waiting periods. To minimize readmission risk, many surgeons prefer in-hospital postoperative monitoring, limiting early discharge.

Recent studies show that connected devices and teleconsultation can provide safe and effective postoperative follow-up. Teleconsultation follow-up is feasible for most patients, with satisfaction rates comparable to in-person visits. Remote monitoring of stoma care has been associated with reduced readmissions. Home-based monitoring using connected vital sign devices in high-risk patients reduces readmissions and emergency visits. In colorectal and bariatric surgery, daily remote monitoring after early discharge (24-48 hours) did not increase morbidity or readmission, suggesting that telemonitoring can safely enable earlier discharge while maintaining patient safety. Continuous monitoring is particularly important for high-risk patients due to rapid deterioration from potential complications.

EPOCA is a telemonitoring and telecoordination platform providing medical, paramedical, and social follow-up at home. It combines connected devices, a digital platform for data analysis, and a dedicated medical and paramedical team. Services include teleconsultations, home paramedical care, support for families or care facilities, and 24/7 emergency management.

EPOCA reassures patients and caregivers, supports primary care and home care teams, and integrates hospital and emergency services. It addresses challenges posed by aging populations, chronic disease prevalence, and increasingly complex patients. By enabling earlier discharge without increasing readmissions, EPOCA offers a holistic solution bridging hospital and home care. It has already demonstrated success in preventing hospitalizations in high-risk elderly patients and is authorized for telemonitoring of chronic conditions including diabetes, respiratory, renal, and cardiac insufficiency.

This study aims to evaluate the feasibility of implementing EPOCA over two years in the CHU Nantes digestive surgery unit. It will target patients undergoing elective or urgent colorectal or bariatric surgery who are at risk of prolonged hospitalization or readmission. High-risk scenarios include anticipated early discharge within 24 hours and patients identified as having elevated readmission risk according to predefined criteria

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age.
* Patients undergoing colorectal or bariatric surgery not routinely managed as outpatient procedures at Nantes University Hospital.
* At least one of the following criteria:
* Anticipated early discharge (within 24 hours post-surgery) for procedures not routinely managed as outpatient at the hospital.
* Estimated risk of readmission greater than 6% according to the Tevis et al. nomogram, adapted to the postoperative context in digestive surgery (>50 points on this score).
* Patients enrolled in a health insurance plan

Exclusion Criteria:

* Discharge to a rehabilitation center requested by the patient
* Condition routinely managed as an outpatient procedure
* Patient under home hospitalization care
* Suicidal or heteroaggressive risk in a patient living alone at home
* Homeless patients
* Pregnant or breastfeeding women
* Patients under legal guardianship, conservatorship, or judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project concerns patients undergoing colorectal or bariatric surgery, either emergent or elective, in the digestive surgery department of Nantes University Hospital, who are at high risk of readmission
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of implementing the EPOCA discharge program in the digestive surgery department of Nantes University Hospital | 90 days post surgery
  Cumulative duration of re-hospitalization days up to 90 days post-surgery (number of day)

SECONDARY OUTCOMES:
Morbidity rate | 90 days
  Postoperative morbidity at 90 days: number of patients experiencing a complication out of the total number of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France